CLINICAL TRIAL: NCT00246597
Title: A Phase III Clinical Trial of PROCRIT (Epoetin Alfa) Versus Placebo in Women Undergoing Adjuvant Chemotherapy for Stage I, II or III Breast Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study stopped to avoid treating enrolled subjects to hemoglobin levels higher than those specified in current labeling.
Sponsor: Ortho Biotech Products, L.P. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002305
Record Dates: First submitted 2005-10-28; First posted 2005-10-31 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-03

CONDITIONS: Anemia; Breast Neoplasms; Hemoglobins; Quality of Life; Chemotherapy, Adjuvant
Keywords: Anemia; Breast cancer; Hemoglobin; Quality of Life; Adjuvant Chemotherapy; Pure red cell aplasia (PRCA); Cognitive and executive function
MeSH Terms: conditions — Anemia; Breast Neoplasms; Red-Cell Aplasia, Pure | interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The purpose of this study is to determine whether it is possible to measure temporary difficulty with thinking and/or short-term memory in women who are receiving chemotherapy for early stage breast cancer and to determine whether or not treatment with PROCRITÂ® will help decrease any problems with thinking or short-term memory that chemotherapy may cause.

DETAILED DESCRIPTION:
Studies of the effect of erythropoietin on rat and mouse brain suggests a neuroprotective and cognitive-enhancing effect of this hormone. The objective of this study was to quantify and compare the incidence of chemotherapy-related impairment of cognitive and executive function in breast cancer patients randomized to receive PROCRIT versus placebo while receiving adjuvant anthracycline-based chemotherapy with or without a Taxane and to evaluate the effect of PROCRIT® on the incidence of asthenia (severe fatigue), quality of life (QoL), and mood. Patients received study medication injections (40,000 units) under their skin once every week for 12 to 24 weeks of chemotherapy. Doses were adjusted depending on the patients' hemoglobin level up to a maximum of 60,000 units.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of Stage I, II or III cancer (chemotherapy naïve for breast cancer) with anthracycline-based adjuvant chemotherapy with or without a taxane
* Hemoglobin >=9 and <=14 g/dL unrelated to transfusion
* Able to read, understand and complete QoL & Cognition tools
* Patients with reproductive potential must have a negative serum pregnancy test within 7 days of study enrollment and use an adequate contraceptive method

Exclusion Criteria:

* Patients who will receive more than a total of 24 weeks of chemotherapy
* psychiatric or neurologic condition that would prevent informed consent and completion of questionnaires or that is poorly controlled with the current treatment regimen
* severe hemiparesis or other condition, distal neuropathy, action tremor or other motor dysfunction, visual deficiencies preventing/decrease bimanual keyboard operation
* severe bradyphrenia (slow thinking) or bradykinesia (slow movement)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2002-12; Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
To assess the effect of PROCRIT® on impairment of cognitive and executive function

SECONDARY OUTCOMES:
To assess the effect of PROCRIT® on severe fatigue, quality of life and mood. Hemoglobin (Hg) Responders were those patients who did not require transfusion during the treatment phase and who demonstrated a > or = 2 g/dL increase in Hg or Hg of 12 g/dL.

CONTACTS AND LOCATIONS:
Overall Officials: Ortho Biotech Products, L.P. Clinical Trial, Study Director — Ortho Biotech Products, L.P.

REFERENCES:
- See also: A Phase III Clinical Trial of PROCRIT� (Epoetin alfa) versus Placebo in Women Undergoing Adjuvant Chemotherapy for Stage I, II or III Breast Cancer — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=921&filename=CR002305_CSR.pdf